CLINICAL TRIAL: NCT04920578
Title: A 3-Part, Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-69095897 in Healthy Participants
Brief Title: A Study of JNJ-69095897 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision to end clinical development of JNJ-69095897
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108935; 2021-000609-26 (EudraCT Number); 69095897EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) Cohorts (Double-blind) (Experimental): Healthy male participants will receive JNJ-69095897 or matching placebo orally in Cohorts 1-8.
  Interventions: Drug: JNJ-69095897; Other: Placebo
- Part 2: Single Dose Cohort (Open-label) (Experimental): Healthy male participants will receive JNJ-69095897 orally in Cohort 9.
  Interventions: Drug: JNJ-69095897
- Part 3: Single or Divided Dose Cohort (Double-blind) (Experimental): Healthy male participants and women of non-childbearing potential (WONCBP) will receive JNJ-69095897 or matching placebo orally in Cohort 10.
  Interventions: Drug: JNJ-69095897; Other: Placebo

INTERVENTIONS:
Drug: JNJ-69095897 — JNJ-69095897 will be administered orally in Parts 1, 2 and 3.
Other: Placebo — Matching placebo will be administered orally in Parts 1 and 3.
  Arms: Part 1: Single Ascending Dose (SAD) Cohorts (Double-blind); Part 3: Single or Divided Dose Cohort (Double-blind)

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-69095897 versus placebo and to characterize the pharmacokinetic (PK) of JNJ-69095897 in blood, plasma, cerebrospinal fluid (CSF) and urine after single or divided oral dose administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise, healthy based on physical examination, medical history, vital signs, orthostatic blood pressure measurements and 12-lead Electrocardiography (ECG) (means of triplicate ECG, inclusive, QT corrected according to Fridericia's formula [QTcF] less than or equal to [<=] 450 millisecond [msec] for males and <= 470 msec for females) performed at screening and admission to the clinical unit. Minor abnormalities in ECG, blood pressure and heart rate, which are not considered to be of clinical significance by the investigator, are acceptable, with the exception of bradycardia <= 45 beats per minutes (bpm) on 12-lead safety ECG, that will be exclusionary at screening, admission to the clinical unit or prior to the first dose on the dosing day
* Otherwise, healthy based on clinical laboratory tests performed at screening. If the results of the serum chemistry panel including liver enzymes, hematology, or urinalysis are outside the normal reference ranges, the participant may be included at the discretion of the investigator, provided the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant has a body mass index (BMI) between 18.0 and 30.0 kilogram/meter square (kg/m^2) inclusive (BMI=weight/height^2)
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for the study and is willing to participate in the study. Participation in the pharmacogenomic part of the study is mandatory

Exclusion Criteria:

* Has a history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other significant cardiac disease, orthostatic hypotension, liver or renal insufficiency, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances or any other illness that the investigator considers should exclude the participant
* Has a diagnosis or suspicions of any sleep disorder in the last 6 months or current complaints of sleep disturbance, irregular sleep schedule or shift work; habitual daytime naps; travel across time zones in the last 4 weeks or daytime symptoms attributable to unsatisfactory sleep
* Has a history of or current major or clinically relevant psychiatric disorder as classified according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) (example, mood, anxiety disorders, psychotic disorder et cetera)
* Has had a clinically significant acute illness within 7 days prior to study intervention administration
* Has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with written concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Vital Sign Abnormalities | Up to Day 14
  Number of participants with vital sign abnormalities including heart/pulse rate, systolic blood pressure, diastolic blood pressure, tympanic body temperature and respiratory rate will be reported.
Number of Participants with Clinical Laboratory Abnormalities (Chemistry, Hematology, Urinalysis) | Up to Day 14
  Number of participants with clinical laboratory abnormalities including chemistry, hematology and urinalysis will be reported.
Number of Participants with Adverse Events (AEs) | Up to Day 14
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 14
  Number of participants with ECG abnormalities will be reported.
Number of Participants with Holter Recording Abnormalities | Up to Day 2
  Number of participants with Holter recording abnormalities (including heart rate variability [HRV]) will be reported.
Plasma Concentration of JNJ-69095897 and its Possible Metabolites | Up to Day 14
  Plasma concentration of JNJ-69095897 and its possible metabolites will be reported.
Part 3: Cerebrospinal Fluid (CSF) Concentration of JNJ-69095897 and its Possible Metabolites | Up to Day 2
  CSF concentration of JNJ-69095897 and its possible metabolites will be reported.
Part 1: Urine Concentration of JNJ-69095897 and its Possible Metabolites | Up to Day 4
  Urine concentration of JNJ-69095897 and its possible metabolites will be reported.

SECONDARY OUTCOMES:
Plasma and CSF Concentration of Endogenous Metabolites | Day 1
  Plasma and CSF concentrations of endogenous metabolites will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jannsen Research & Development, LLC Clinical Trial, Study Director — Jannsen Research & Development, LLC
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency